CLINICAL TRIAL: NCT03731767
Title: The Effect of a Talocrural Thrust Manipulation on Lateral Ankle Ligament Integrity in a Subgroup of Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FloridaGCU 2018-50
Record Dates: First submitted 2018-10-29; First posted 2018-11-06 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Manipulation; Thrust; Ankle; Ligaments

STUDY DESIGN:
Intervention Model Description: Pretest post test study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject group (Other): Distraction thrust manipulation of the talocural joint in supine position
  Interventions: Procedure: Distraction thrust manipulation

INTERVENTIONS:
Procedure: Distraction thrust manipulation — Distraction thrust manipulation of the talocural joint in supine position

SUMMARY:
Measure the effect of a common used ankle manipulation on ligament length in the ankle.

DETAILED DESCRIPTION:
The purpose of this study is to determine what the effect of a common ankle manipulation on the supporting ligaments of the ankle.

Design: The researchers will conduct a quasi-experimental study with a method of convenience sampling. The design of this study will allow to determine what the direct effect of a common a commonly used physical therapy ankle manipulation is on the length of the soft tissue connection between the smaller bone in the lower leg and the heel bone and the smaller bone in the leg and the ankle bone.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years old
2. No current trauma to the ankle/ foot-if not present both ankles will be used during this study
3. No hx of fracture or surgical intervention to the ankle

Exclusion Criteria:

1. Red flags identified during the subjects intake. If manipulation is contraindicated the subjects will be removed from the study.
2. History of ankle/ foot trauma within the last 3 months.
3. History of surgery on the ankle/ foot.
4. History of knee, hip, or lower back related issues that would make the application of the ankle manipulation contraindicated.
5. Workers compensation and any pending legal action regarding ankle/ foot related issues.
6. Undergone any ankle manipulation within the last 3 weeks.
7. History of Osteopenia or Osteoporosis.
8. Inability to undergo measuring protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Tendon length | Measure 1 prior to manipulation. Measure 2 immediately after manipulation, within 5 minutes (the same day)
  Change in ankle ligament length in millimeters measured by a method of musculoskeletal Ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, Principal Investigator — FGCU Assistent Professor
Locations (1):
- Integrated Therapy Practice PC, Cape Coral, Florida, United States

IPD SHARING:
Plan to Share IPD: No